CLINICAL TRIAL: NCT03134183
Title: A Randomized Double-blinded Comparison of 24-hour Interval-Mifepristone and Buccal Misoprostol Versus Mifepristone and Vaginal Misoprostol for Cervical Preparation in Second-Trimester Surgical Abortion
Brief Title: 24-hour Mifepristone and Buccal Versus Mifepristone and Vaginal Misoprostol for Cervical Preparation for D&E
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HM20005740
Record Dates: First submitted 2017-04-25; First posted 2017-04-28 (Actual); Results first posted 2018-07-18 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-06

CONDITIONS: Abortion, Second Trimester
Keywords: D&E; dilation and evacuation; abortion; second trimester; mifepristone; misoprostol
MeSH Terms: conditions — Dilatation, Pathologic | interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Computer-generated randomization will be utilized to assign treatment arms and the vaginal misoprostol and buccal placebo and buccal misoprostol and vaginal placebo will be prepared according to randomization scheme by the research pharmacy in opaque-sealed envelopes as to blind participants and providers.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vaginal Misoprostol (Experimental): Intervention is misoprostol versus placebo 400mcg misoprostol formulated within cocoa butter suppository
  Interventions: Drug: Vaginal Misoprostol
- Buccal Misoprostol (Experimental): Intervention is misoprostol versus placebo 400mcg misoprostol formulated within mint flavored powder
  Interventions: Drug: Buccal Misoprostol

INTERVENTIONS:
Drug: Vaginal Misoprostol — Mifepristone 200mg orally 20-24 hours prior and misoprostol 400mcg (two 200mcg tablets) vaginally 1-2 hours prior and placebo (buccal mint powder) buccally 1-2 hours prior to D&E
  Other Names: cytotec
  Arms: Vaginal Misoprostol
Drug: Buccal Misoprostol — Mifepristone 200mg orally 20-24 hours prior and misoprostol 400mcg (two 200mcg tablets) ground with mint into buccal powder and placebo (two lactose tablets designed to appear similar to misoprostol) vaginally 1-2 hours prior to D&E
  Other Names: cytotec
  Arms: Buccal Misoprostol

SUMMARY:
This study aims to compare mifepristone and buccal misoprostol to mifepristone and vaginal misoprostol for cervical preparation for second trimester dilation and evacuation (D&E).

DETAILED DESCRIPTION:
Standard of care for cervical preparation prior to second trimester surgical abortion has traditionally been a pelvic exam with speculum, a paracervical block with lidocaine, and placement of a number of osmotic dilators through the cervical canal. Dilators obtain maximal expansion within 4-6 hours and patients experience cramping with this process. This cervical preparation allows for a faster procedure for the patient (limiting time for anesthesia) and an easier procedure for the provider (decreasing necessity for further dilation, decreasing risk of cervical laceration, and decreasing blood loss). Following cervical preparation, trained providers use instruments to remove the pregnancy per standard of care. Several studies have examined the use of medication (mifepristone and/or misoprostol) to dilate the cervix as an alternative to osmotic dilators . Patients prefer medication to dilators as medication is associated with less discomfort. Medications alone can achieve adequate cervical preparation but the optimal timing and routes of these medications has not been sufficiently evaluated.

The addition of mifepristone, a progesterone antagonist, to a misoprostol regimen has been shown to significantly decrease the medication-to-abortion interval in second-trimester induction terminations. Vaginal administration has demonstrated improved dilation as compared to buccal administration but it is known that patients prefer buccal administration. A comparison of mifepristone and vaginal versus mifepristone and buccal misoprostol has not been studied prior to second-trimester surgical abortion.

A review of cervical preparation for second-trimester D&E did not recommend mifepristone and misoprostol for cervical priming due to high rates of pre-procedural expulsions. However, the primary basis for this conclusion is a trial in which the 48-hour interval between the medications accounts for the high out-of-facility expulsion risk. A retrospective cohort of over 200 women between 14 and 19 6/7 weeks gestation showed no difference in difficulty of cervical dilation for patients receiving mifepristone 24-48 hours misoprostol as compared to osmotic dilators prior to surgical abortion. Two out of facility expulsions occurred in the mifepristone-misoprostol arms but the timing of medication to expulsion interval is not reported.

More recent studies have limited the timing of mifepristone to 24 hours or less prior to procedure. Mifepristone only has been shown to provide adequate cervical dilation as compared to osmotic dilators to 16 weeks gestation with noninferiority design to detect a 3-minute difference in procedure time. A 24-hour interval between 200mg mifepristone and 400mcg buccal misoprostol has been shown as non-inferior to osmotic dilators for total procedure time for 15-18 week surgical abortions. Mifepristone and one-set of osmotic dilators was found to be non-inferior for total procedure time as compared to two sets of osmotic dilators for surgical abortion 19-23 6/7 weeks gestation.

The addition of mifepristone has benefit as a cervical priming agent as an adjunct or alternative to osmotic dilators for surgical abortion, but it is not known whether the addition of vaginal versus buccal misoprostol changes cervical dilation and thus procedure time outcomes.

ELIGIBILITY:
Inclusion Criteria:

* The study will enroll healthy English or Spanish-speaking women, over 18 years of age, eligible for non-urgent D&E at 16 0/7 weeks to 20 6/7 weeks gestation, confirmed by sonogram, and willing/able to undergo informed consent.

Exclusion Criteria:

* Emergent need for D&E, intrauterine infection, fetal demise, molar pregnancy, intolerance, allergy or contraindication to mifepristone or misoprostol

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2016-11-19 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frances Casey, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vaginal Misoprostol | Buccal Misoprostol
Started | 36 | 34
Completed | 35 | 33
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vaginal Misoprostol | Buccal Misoprostol | Total
Number analyzed (Participants) | 35 | 33 | 68
Age, Customized [Count of Participants; unit: Participants]
  18-24 | 13 | 16 | 29
  25-29 | 9 | 6 | 15
  30-34 | 4 | 7 | 11
  35+ | 10 | 5 | 15
Sex: Female, Male [Count of Participants; unit: Participants] — Men not eligible for study. N/A
  Participants
    Female | 35 | 33 | 68
    Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 35 | 33 | 68

OUTCOME MEASURES:

1. Primary Outcome: Procedure Time
Description: Time from initial uterine instrumentation to speculum out
Time Frame: At end of procedure
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Vaginal Misoprostol | Buccal Misoprostol
Number analyzed (Participants) | 35 | 33
minutes | 9.5 (5) | 9.9 (4)

2. Secondary Outcome: Cervical Dilation
Description: Pratt Dilator initially accepted without resistance starting from 65 and working down
Time Frame: At end of procedure
Measure: Mean (Standard Deviation); unit: "French" circumference in millimeters
Arm/Group | Vaginal Misoprostol | Buccal Misoprostol
Number analyzed (Participants) | 35 | 33
"French" circumference in millimeters | 49.6 (10) | 46.2 (11)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Vaginal Misoprostol | Buccal Misoprostol
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/33
Other Adverse Events (participants affected / at risk) | 1/36 | 0/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaginal Misoprostol (N=36) | Buccal Misoprostol (N=34)
Expulsion (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-15): https://cdn.clinicaltrials.gov/large-docs/83/NCT03134183/Prot_SAP_000.pdf